CLINICAL TRIAL: NCT00936169
Title: Angiography vs. IVUS Optimisation: A Multi-Centre European Study of Drug Eluting Stent Implantation
Brief Title: Angiography Versus (vs) IVUS Optimisation
Acronym: AVIO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Evidence per Attività e Ricerche Cardiovascolari ONLUS (Other)
Collaborators: Mediolanum Cardio Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AVIO
Record Dates: First submitted 2009-07-08; First posted 2009-07-09 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2009-07

CONDITIONS: Myocardial Infarction
Keywords: Patients with at least one complex lesion suitable for implantation of a drug-eluting stent
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IVUS optimised stent implantation (Experimental)
  Interventions: Procedure: IVUS optimised DES implantation
- angiographically guided DES implantation (Active Comparator)
  Interventions: Procedure: angiographically guided DES implantation

INTERVENTIONS:
Procedure: IVUS optimised DES implantation — Ivus optimised stent implantation
  Arms: IVUS optimised stent implantation
Procedure: angiographically guided DES implantation — angiographically guided DES implantation
  Arms: angiographically guided DES implantation

SUMMARY:
The purpose of the study id to demonstrate an advantage for intra-vascular ultrasound (IVUS) optimized drug-eluting stent (DES) implantation compared to angiography in complex lesions

ELIGIBILITY:
Inclusion Criteria:

* A complex lesion is regarded as a lesion where the operator would expect a lower immediate and long term success rate compared to non-complex lesions (according to the results of Randomized Controlled Trials and from large Registries). The operator must consider the implantation of a drug-eluting stent, feasible and appropriate for this particular complex lesion

Exclusion Criteria:

* Contra-indication to dual anti-platelet therapy.
* Ejection fraction <30%.
* Renal failure (creatinine >2 mg/dL).
* Significant co-morbidity precluding clinical follow-up.
* Acute myocardial infarction in the 48 hours prior to the procedure.
* In-stent restenosis
* Prior brachytherapy
* Thrombocytopenia <100,000
* Unprotected left main stem stenosis
* Venous or arterial grafts
* Recipient of heart transplant
* A positive pregnancy test in women with child bearing potential
* Acute infections
* Major surgery planned which will lead to discontinuation of antiplatelet therapy
* Patients with prior BMS or DES implanted in the target vessel less than one year prior to the enrollment, including one year from any intercurrent restenotic or thrombotic event
* Age under 18 years old.
* There is no maximum number of lesions which can be treated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 284 (Actual)
Dates: Start 2008-05; Primary Completion 2009-06 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Post-procedure Minimal Lumen Diameter (MLD) evaluated by core lab QCA: superiority for the IVUS optimised group. | Procedure day

SECONDARY OUTCOMES:
Target lesion revascularisation (TLR) at 9 months: superiority or statistical trend for the IVUS optimized group | 9 months
Major adverse cardiac events (MACE) at 9 months: superiority or statistical trend for the IVUS guided group due to lower TLR and no difference in myocardial infarction (MI) or death. | 9 months
MACE events at 2 years. | 2 years

REFERENCES:
- [Derived] Chieffo A, Latib A, Caussin C, Presbitero P, Galli S, Menozzi A, Varbella F, Mauri F, Valgimigli M, Arampatzis C, Sabate M, Erglis A, Reimers B, Airoldi F, Laine M, Palop RL, Mikhail G, Maccarthy P, Romeo F, Colombo A. A prospective, randomized trial of intravascular-ultrasound guided compared to angiography guided stent implantation in complex coronary lesions: the AVIO trial. Am Heart J. 2013 Jan;165(1):65-72. doi: 10.1016/j.ahj.2012.09.017. Epub 2012 Nov 20. PMID 23237135